CLINICAL TRIAL: NCT02758535
Title: Renal Parenchymal Core Needle Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modarres Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Renal Parenchymal Biopsy
Record Dates: First submitted 2016-04-29; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Image-guided Biopsy; Complications; Kidney Glomerulus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Core needle biopsy with coaxial method (Experimental): The patients undergo renal biopsy with a coaxial Tru-Cut needle
  Interventions: Device: coaxial renal biopsy
- Core needle biopsy with noncoaxial method (Experimental): The patients undergo renal biopsy with a noncoaxial Tru-Cut needle
  Interventions: Device: noncoaxial renal biopsy

INTERVENTIONS:
Device: coaxial renal biopsy — In this method, a larger introducing needle is used for the puncture. The introducing needle is advanced just to the outer cortex of the kidney, and the needle angle is adjusted so that the needle pathway became mostly in the renal cortex, then the biopsy needle is inserted throughout the introducing needle and at least 4 cores are obtained. In this technique, the skin surface is punctured only once during the procedure.
  Other Names: 18-gauge semiautomatic biopsy system with the coaxial needle; Tasuku Laboratory, Tochigi, Japan
  Arms: Core needle biopsy with coaxial method
Device: noncoaxial renal biopsy — In this method, introducing needle is not used. Biopsy needle punctures the skin surface and the needle is advanced to about 10-15 mm into the renal cortex, and tissue sampling is done. After each sampling, the needle is removed and then for the next biopsy, the whole procedure is repeated until four cores being taken.
  Other Names: 18-gauge semiautomatic biopsy system without coaxial needle; Tasuku Laboratory, Tochigi, Japan
  Arms: Core needle biopsy with noncoaxial method

SUMMARY:
Percutaneous image-guided parenchymal renal biopsy has been used to detect the different pathologies of renal parenchyma, to define the degree of reversible changes, and to define when the medical treatment fails. Percutaneous core needle renal biopsy has been reported to have a higher diagnostic yield compared to fine needle aspiration. Percutaneous core needle renal biopsy is usually based on tissue sampling under guidance of either sonography or computed tomography. Renal parenchymal biopsy can be done either with a coaxial or noncoaxial technique. In coaxial technique, the introducing needle is placed in the renal parenchyma; then, multiple tissue sampling can be performed throughout the same tract. Alternatively, in noncoaxial technique, biopsy needle is inserted repeatedly for each tissue sampling. Although there are some reports regarding the comparison of coaxial and noncoaxial methods of renal mass biopsy, comparison of the two methods in renal parenchymal biopsy has not yet been described in the literature. In this prospective study, the investigators sought to compare the procedural time and the complication rate of coaxial technique with those of noncoaxial technique in percutaneous renal parenchymal biopsy.

ELIGIBILITY:
Inclusion Criteria:

* impaired renal function
* proteinuria
* hematuria

Exclusion Criteria:

* renal hydronephrosis
* chronic renal failure
* a history of renal cell carcinoma
* suspicious renal mass
* uncorrectable coagulopathy

Ages: 10 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
complication ratio | within 48 hours after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Poursina Hospital, Guilan University of Medical Sciences, Rasht, Gilan Province, Iran

IPD SHARING:
Plan to Share IPD: No